CLINICAL TRIAL: NCT00826605
Title: Retrospective Investigation of Presence of Urobilinogen and Maternal Weight Loss as Indications of Impending Parturition in the Term Gravida
Brief Title: Urobilinogen, Maternal Weight Loss and Impending Parturition at Term
Status: Completed | Type: Observational
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Elizabeth Harris, DO, OB/Gyn Resident, Oklahoma State University Center for Health Sciences
Other Study IDs: 200802
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Increase in Urobilinogen in Urine Prior to Delivery; Weight Loss After 37 Weeks Gestation Prior to Delivery
Keywords: Weight loss, urobilinogen
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Urobilinogen increase: Increase in urobilinogen increase on routine dipstick test at prenatal appointment after 37 weeks gestation
- Weight Loss at Term: Weight loss since previous prenatal appointment after 37 weeks gestation

SUMMARY:
The purpose of this study, then, is to search existing clinic and hospital records for answers to the following two questions: (1) Do pregnant women who are at least 37 weeks gestation and who have an increase in urubilinogen on urine dipstick at a prenatal appointment have a statistically significant shorter average time before going into active labor than their negative counterparts? (2) Do pregnant women who are at least 37 weeks gestation and who show a modest weight loss between two prenatal appointments have a statistically significant shorter average time before going into active labor than their counterparts who did not lose weight?

DETAILED DESCRIPTION:
Rationale/Background:

This study is a retrospective review of records which examines the possibility of two markers for the onset of active labor (contractions which result in a change in the uterine cervical dilatation) on routine clinical prenatal assessment. The markers in question are an elevation of urobilinogen on routine dipstick and slight maternal weight loss. An apparent clinical correlation between the presence of urobilinogen, maternal weight loss and onset of active labor has been observed in our patient population. Our hypothesis is that these markers in the term gravida are an indication of delivery within a week of their appearance on routine prenatal evaluation. Should a correlation exist, the clinician would have a relatively inexpensive way of identifying patients that could deliver within the week and could possibly predict those patients that would have success with induction, as the normal labor process may have begun. The purpose of this study, then, is to search existing clinic and hospital records for answers to the following two questions: (1) Do pregnant women who are at least 37 weeks gestation and who have an increase in urobilinogen on urine dipstick at a prenatal appointment have a statistically significant shorter average time before going into active labor than their negative counterparts? (2) Do pregnant women who are at least 37 weeks gestation and who show a modest weight loss between two prenatal appointments have a statistically significant shorter average time before going into active labor than their counterparts who did not lose weight? In humans, the signals that initiate labor are not completely understood. While many theories have been explored, an exact pathway has not yet been determined. Urobilinogen is formed from conversion of conjugated bilirubin in the intestine by bacteria. A fraction of the urobiliogen is then reabsorbed into the bloodstream and filtered by the kidneys, becoming a colorless component of urine. Normally, only 1-4 mg of urobilinogen is excreted in the urine per day. Hemolytic processes, hepatocellular damage, and cholestasis can elevate urobilinogen in the urine. Routine dipstick tests have a normal urobilinogen range of 0.2 to 1 mg/dl (1). In this study, we will examine the urine dipsticks for an increased change in the urobilinogen levels within the last two prenatal appointments prior to delivery.

No previous studies could be located regarding a link between an elevation in urobilinogen and/or minor maternal weight loss and parturition, labor, onset. There have been studies to suggest rationale for our clinical observation, however. Estrogens and progesterone both play a role in the growth and contractility of uterine myometrial cells. Progesterone tends to promote uterine relaxation, hence the name "pro-gest…". In most species, progesterone levels dramatically fall, a 'withdrawal', prior to the onset of labor. However, in human and higher level primates, the progesterone and estrogen levels are both elevated in later gestation and during parturition. The "withdrawal" in humans, therefore, may be mediated by changes in the myometrial responsiveness to progesterone (2).

Estrogens induce myometrial contractility. Estriol is the most abundant estrogen during pregnancy and is produced by the placenta. It first appears at approximately the ninth week of gestation from the last menstrual period (3). Plasma concentrations of this estrogen increase throughout gestation along with those of estrone and estradiol (3,4,5). In the weeks preceding parturition, concentrations of estriol dramatically increase and continue to rise until birth (6). Estriol's roles include preparing uterine tissues for contraction and possibly signaling parturition in higher primates and humans (3,4,7,8,9,10). A rise in estriol, which can be monitored in saliva, has been shown to precede parturition, regardless of whether labor begins preterm, at term, or postterm (11,12).

Estrogens' effect on the liver has been studied extensively. The active transport of biliary components in the canaliculi is impaired by estrogen (13). The pregnant state can cause some changes in bile acid production and secretion, presumably due to the higher levels of estrogen, but also because of progesterone's effect on GI motility. This can lead to a mild subclinical cholestasis. Studies have shown conflicting evidence as to whether there is an increase in bile acid levels during pregnancy. As estrogen increases are known to induce a cholestasis, and urobilinogen levels increase in cholestasis, our hypothesis is that the increase in estrogen levels within the last week of pregnancy may slow the clearance of bile even further yielding the rise in urobilinogen levels noticed on routine dipstick.

An in depth literature review was performed in an effort to find a correlation between maternal weight loss and the onset of labor. No supporting literature validated or explained our clinical observation.

Methodology This study will be a retrospective chart review of all eligible patients who presented to labor and delivery at Oklahoma State University Medical Center between the dates of January 1, 2002 and December 31, 2006. We selected this particular time period of charts to review, because they are recent enough to be accessible, and we estimate they will yield usable data for about 200 women.

The study population will include mothers between the ages of 18 and 34 years of age with a single intrauterine pregnancy between 37 weeks and 41 weeks gestational age. (Both very young mothers and women 35 and older have increased risk of premature delivery.) The patients will have an admission diagnosis of either active labor or spontaneous rupture of membranes. Active labor is defined as uterine contractions resulting in changes either in the cervical dilatation, the effacement of the cervix and/or descent of the fetal head in the pelvis.

This study will review chart data collected from our obstetrical clinic, OSU Obstetrics and Gynecology, as well as OSU Medical Center records. We will first search the hospital's records for patients admitted with the diagnosis of active labor. These charts will be examined for inclusion/exclusion criteria and entered into the study if they are eligible (as later defined). Once these charts have been obtained, we will then search their corresponding clinic chart for the defined parameters of our study.

Eligibility Criteria:

Our study population will consist of women between the ages of 18 and 34 who delivered a single, viable, term infant at OSU Medical Center between January 1, 2002 and December 31, 2006. Gestational age must be greater than 37 weeks and less than 41 weeks, as ascertained by certain last menstrual period and/or first trimester ultrasound. The chart must include a diagnosis of active labor or spontaneous rupture of membranes, and the patient must have had at least two third-trimester prenatal checkups at OSU Houston Center OB/GYN, including one during the last two weeks of gestation. We will define a term infant as 37 weeks gestation or greater (3). Our study population will consist of mainly Medicaid patients. The ethnic blend of our study population will include Caucasian, African-American, Hispanic, American Indian, and Asian women.

We will exclude women with multiple gestation, because they are at risk of preterm labor. We will also exclude anyone else who had preterm delivery. In addition, we will exclude women with a diagnosis of liver disease, including intrahepatic cholestasis and hepatitis, chronic hypertension, intraamniotic infection, preeclampsia or its variant, HELLP syndrome, cholelithiasis, inadequate prenatal care, preterm labor, or induction of labor (other than due to premature rupture of membranes).

Data Collection Only the investigators will have access to the patients' data collection sheet. Individual physicians involved in the care of a specific patient will have access to that patient's information. All individuals will be in compliance with HIPPA guidelines as set forth by the university and the medical center. Patient records will be locked in a file cabinet or kept with their regular charts in the patient records department of the OSU Houston Center OB/GYN clinic. Any information obtained from hospital labor and delivery charts will be collected by Dr. Harris. It will be directly transported from the hospital to the clinic only by her, will be kept on her person at all times en route, and will be stored in a locked folder while in transit.

The following data will be collected from the patients' hospital record.

1. Name
2. Birthdate
3. Age of patient (years)
4. Medical Record Number (MRN)
5. Gestational age (in weeks and days)/Determined by:
6. Initial sterile vaginal exam results (normal yes/no)
7. Date and time of admission
8. Admission Diagnosis
9. Date and time of delivery
10. Co-morbidities, pregnancy complications
11. Delivery Mode
12. Indication for Cesarean Section if applicable Note that it is not possible to determine the time of onset of active labor, only the time of hospital admission. We are assuming that most women who go into active, natural labor present to the hospital within 12-18 hours. The day of hospital admission, then, serves as a rough, best estimate for onset of natural, active labor.

The following data will be collected from the patients' clinic record.

1. Patient's Name
2. Birthdate
3. Age
4. MRN (megawest number)
5. Date of delivery (from hospital record)
6. Date of first clinic visit
7. Number of clinic visits
8. Weight on first clinic visit
9. Total pregnancy weight gain
10. Date of last clinic visit
11. Weight at that visit
12. Urine dipstick result at that visit
13. Sterile vaginal exam (SVE) (dilation, effacement, station) at that visit
14. Date of Visit prior to last clinic visit
15. Weight at that visit
16. Urine dipstick result at that visit
17. SVE at that visit
18. Pregnancy Complications

Note that after 36 weeks gestation, prenatal visits are scheduled weekly at OSU Clinics. Therefore, unless the patient is not compliant with routine visits, natural labor for a term pregnancy will take place no longer than seven days from last clinic visit. No other data will be collected from any patient charts.

Analysis:

Data will be analyzed using PC SAS Version 9.1 (SAS Institute, Cary, NC). The two components of the study will be analyzed separately. The weight loss leg of the study will utilize an independent t-test in an effort to determine the relationship of weight loss (yes/no) to time to delivery. For the urobilinogen component of the study, we will utilize correlation techniques to assess the relationship of time to delivery and urobilinogen level. Significance will be determined at the 0.05 level.

Confidentiality:

All records and lab results will be maintained at Oklahoma State University Medical Center, department of medical records and laboratory storage on the hospital's Meditech system. All of the documents linking patient names to these numbers and charts will be destroyed after data collection is complete.

ELIGIBILITY:
Inclusion Criteria: Our study population will consist of women between the ages of 18 and 34 who delivered a single, viable, term infant at OSU Medical Center between January 1, 2002 and December 31, 2006. Gestational age must be greater than 37 weeks and less than 41 weeks, as ascertained by certain last menstrual period and/or first trimester ultrasound. The chart must include a diagnosis of active labor or spontaneous rupture of membranes, and the patient must have had at least two third-trimester prenatal checkups at OSU Houston Center OB/GYN, including one during the last two weeks of gestation. We will define a term infant as 37 weeks gestation or greater (3). Our study population will consist of mainly Medicaid patients. The ethnic blend of our study population will include Caucasian, African-American, Hispanic, American Indian, and Asian women.

-

Exclusion Criteria: We will exclude women with multiple gestation, because they are at risk of preterm labor. We will also exclude anyone else who had preterm delivery. In addition, we will exclude women with a diagnosis of liver disease, including intrahepatic cholestasis and hepatitis, chronic hypertension, intraamniotic infection, preeclampsia or its variant, HELLP syndrome, cholelithiasis, inadequate prenatal care, preterm labor, or induction of labor (other than due to premature rupture of membranes).

-

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Population is mothers between the ages of 18 and 34 years of age with a single intrauterine pregnancy between 37 weeks and 41 weeks gestational age. (Both very young mothers and women 35 and older have increased risk of premature delivery.) The patients will have an admission diagnosis of either active labor or spontaneous rupture of membranes. Active labor is defined as uterine contractions resulting in changes either in the cervical dilatation, the effacement of the cervix and/or descent of the fetal head in the pelvis.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Increase in urobilinogen on routine urine dipstick at prenatal appointment, term pregnancy | none--chart review

SECONDARY OUTCOMES:
Maternal weight loss at term before giving birth | none--chart review

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Harris, DO, Principal Investigator — OSU Center for Health Sciences
Locations (2):
- United States (2):
  - OSU Houston Center OB/Gyn Clinic, Tulsa, Oklahoma
  - OSU Medical Center, Tulsa, Oklahoma